CLINICAL TRIAL: NCT07185568
Title: IntraOperative UltraSound Guided Versus Wire Guided Versus Magnetic Seed Guided Breast-conserving Surgery for Non-palpable Tumors.The MANOLA Study Multi-center, Randomized, Open-label Clinical Trial
Brief Title: IntraOperative UltraSound Guided vs Wire Guided vs Magnetic Seed Guided Breast-Conserving Surgery for Non-palpable Tumors
Acronym: MANOLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IOV-BC-1-2024 MANOLA
Record Dates: First submitted 2025-09-05; First posted 2025-09-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Breast-Conserving Surgery
Keywords: IntraOperative UltraSound guided; Wire guided; Magnetic Seed guided
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a multi-center, randomized, open-label clinical trial that will enroll 1302 adult patients with non-palpable breast lesions. Participant eligible for the study will be randomized in a 1:1:1 ratio to one of the pre-surgery lesion localization: IOUS HydroMark™ (experimental arm A), magnetic Sirius Pintuition Seed® (experimental arm B) and the wire localization technique (control arm).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IntraOperative Ultrasound (IOUS) HydroMark™ (Experimental): It is an advanced localization technique for non-palpable breast lesions, leveraging real-time ultrasound guidance combined with an ultrasound-visible tissue marker (HydroMark™) to facilitate precise tumor resection during breast-conserving surgery (BCS).
  Interventions: Procedure: IOUS HydroMark™
- Magnetic Sirius Pintuition Seed® (Experimental): It is an advanced, wire-free localization system designed for precise surgical guidance in non-palpable breast lesions. This technology utilizes a small, permanent magnetic seed that can be implanted into the tumor days, weeks, or even months before surgery, offering greater flexibility compared to traditional wire localization.
  Interventions: Procedure: Magnetic Sirius Pintuition Seed®
- Wire localization (Active Comparator): It is the most widely used preoperative technique for guiding the surgical removal of non-palpable breast lesions. This method involves the insertion of a thin hooked wire into the lesion under radiological guidance (ultrasound, mammography, or stereotactic guidance) on the day of surgery. The wire serves as a physical guide for the surgeon, ensuring precise excision of the target lesion.
  Interventions: Procedure: Wire localization (WL)

INTERVENTIONS:
Procedure: IOUS HydroMark™ — IOUS HydroMarkTM allows marking the tissue during percutaneous breast biopsy. This is a sterile, single-use marker made of resorbable hydrogel, which expands upon contact with bodily fluids and is then gradually absorbed. The hydrogel is visible on ultrasound. Inside the hydrogel, there is a metallic spiral (titanium/steel) that remains permanently visible in radiographic and MRI examinations even after the hydrogel has been fully absorbed.
  The HydroMARK Breast Biopsy Site Marker is made of a resorbable hydrogel that expands with fluid and is then resorbed. The hydrogel material is visible under ultrasound. Embedded in the hydrogel is a coiled metallic wire that will be permanently visible under x-ray and MRI when the hydrogel is resorbed. The HydroMARK Biopsy Site Marker is a permanent implant and is not intended to be removed unless the marked tissue is determined to require surgical removal. The marker is supplied pre-loaded in applicator devices designed.
  Arms: IntraOperative Ultrasound (IOUS) HydroMark™
Procedure: Magnetic Sirius Pintuition Seed® — The Pintuition Localization System is intended as a magnetic soft tissue localization system.
  The magnetic Pintuition Seed is indicated for preoperative percutaneous implantation into soft tissue (glandular, fibrous or fatty tissue of breast; lymph nodes in the axillary and inguinal region; subcutaneous tissue and skeletal muscle tissue) for temporary marking (<180 days) of a tissue of interest (e.g. tumor or a suspected lesion) indicated for surgical removal. Using the Pintuition Detector as magnetic guidance or, alternatively, image guidance (ultrasound or x-ray), the Pintuition Seed can be intra-operatively localized and removed together with the tissue of interest.
  Arms: Magnetic Sirius Pintuition Seed®
Procedure: Wire localization (WL) — Single-use, repositionable needle for preoperative localization of breast nodules with a single hook, equipped with a depth limiter. Designed for the localization of non-palpable breast lesions in the preoperative phase. It includes a fixation clamp to stabilize the positioning of the wire.
  Arms: Wire localization

SUMMARY:
This is a multi-center, randomized, open-label clinical trial that will enroll 1302 adult patients with non-palpable breast lesions. Participant eligible for the study will be randomized in a 1:1:1 ratio to one of the pre-surgery lesion localization: IOUS HydroMark™ (experimental arm A), magnetic Sirius Pintuition Seed® (experimental arm B) and the wire localization technique (control arm). The randomization will be stratified by lesion type (solid non-palpable (type B); non-solid non-palpable (e.g., microcalcification clusters, architectural distortive areas) (type C); post-NACT residual lesions (type D), and clinical center.

DETAILED DESCRIPTION:
Breast-conserving surgery is the gold standard treatment for early breast cancer, since it has shown disease-free survival rates equivalent to those of mastectomy, offering the advantages of cosmetic outcome preservation, a better quality of life and a decrease in psychological morbidities. These important aspects, along with the general goal of reducing the extent of surgical excisions, have increased the need for an effective pre- surgery lesion localization and surgical guidance techniques. Reported rates of margin involvement after BCS range from 10 to over 40%, and positive resection margin is one of the strongest predictive factors for local recurrence. This event requires additional surgical procedures (re-excision or mastectomy) and/or radiotherapy boost, leading to higher healthcare costs and worse cosmetic outcomes, in addition to further stress for surgeons and patients.

Wire localization (WL) is the most used method for non-palpable breast lesions, with clear margins reported in a range of 70.8%-87.4% of cases. Recognized advantages of wires are the widespread availability and the moderate price. Moreover, wires emit no ionizing radiation and can be stored safely. Although WL is highly effective, with approximately 2.5% of unsuccessful wire localizations associated with multiple lesions, small lesions, lesions containing extensive microcalcifications and small surgical specimens, it still yields several disadvantages. The procedure is unpleasant and causes patient discomfort; wire migration within the breast, and more infrequently outside the breast, has also been reported. The hookwire can be transected during the surgery, with pieces being retained in the breast post- operatively. Finally, this localization approach requires adequate coordination between trained breast radiologists and surgeons because the wire placement has to occur on the day of surgery to avoid displacement. This limitation can lead to inconvenience and delay in the operating room or suboptimal localization. Moreover, wire localization could limit the surgical approach and cause a potential worse cosmetic outcome; the placement route of the wire, chosen by the radiologist, often dictates incision choice for the surgeon who then has to follow the wire's course during dissection.

Magnetic seed is a relatively new localization technology for non-palpable breast lesions. The localization system includes a magnetic seed, that may be positioned using a needle under radiological guidance days, weeks or months before the surgical procedure and it offers a demonstrated reduced risk of migration compared to wire-guided localization. This method has no radiation emission, so that the signal does not decay over time, and it does not require a destruction protocol in comparison to radioactive seeds. Literature describes magnetic guidance as safe and feasible. The magnetic seeds may be seen on breast imaging including ultrasound, mammography, and tomosynthesis. MRI is not contraindicated although a degree of movement artifact would be expected as with any metal clip. The magnetic device has the potential of localizing lesions accurately, and may reduce re- excision rates, pain and excision specimen weight. The main disadvantages of magnetic seed are the high costs of devices and the creation of MRI artefacts. Nevertheless, magnetic seed localization still seems to be one of the most promising recent technological innovation in BCS. The Sirius Pintuition Seed® is a permanent magnetic seed that accurately marks the tumor and helps the procedure of surgical removal from any direction. The magnetic seed is robust and is encapsulated in high-grade, nickle-free biocompatible titanium. Sirius Pintuition is a wire-free localization technology designed to provide navigational guidance through a dedicated software that offers directional guidance using audio and visual feedback.

All the traditional breast localization techniques may be described as essentially blind, since they do not allow the direct visualization of breast lesions during surgery. In 1988 Rifkin et al. firstly described ultrasound (US) as a tool for localizing breast masses during surgery and facilitating their surgical excision. Many other successful experiences followed, for palpable and non-palpable BC and even for post neoadjuvant residual lesions. A recently published prospective study demonstrated the efficacy of IOUS for all the types of BC lesions. Nevertheless, systematic US performance during BCS is still regarded as a new developing concept, being underused in this surgical oncology field. Intra-operative ultrasound-guided surgery (IOUS) is the only technique allowing a real-time visualization of BC and resection margins running control during all surgical phases. Previous series reported glaring advantages over the other techniques both for oncological and cosmetic outcomes.

HydroMarkTM clip has the potential to amplify the efficacy of IOUS, since the clip is easy to view, and it allows an easier guide in every phase of surgery. The HydroMarkTM marker hydrogel hydrates to provide up to 12 months of ultrasound visibility and it offers permanent stereotactic, tomosynthesis, and X-ray visibility. Moreover, it does not contraindicate Magnetic Resonance Imaging (MRI). It is demonstrated that the clip offers a permanent MRI visibility without generating any artefact, while it results uniquely distinguishable on a T2 sequence for up to 12 months. The results of a recently published study described the procedure of localization the clip under ultrasound as a faster and more comfortable procedure for the patient compared to the wire localization. HydroMark clip costs are slightly higher than a stadard stereotactic clip. The use of IOUS with HydroMark clips have the potential to improve patients' experience, with a particular attention in preserving the cosmetic aspect, leading to an improved quality of life in this specific population. According to the available scientific evidences IOUS technique allows excellent oncological and cosmetic outcomes and contribute to organizational aspects improvement in breast-conserving surgery compared with the traditional methods of wire-guide surgery. Moreover, it seems to be cost-saving with respect to magnetic seeds techniques, without limiting the possibility of further MRI evaluations of the patients.

However only limited literature is available and clinical studies to evaluate safety and effectiveness involving these devices have been carried out on small numbers of patients and not randomized. No strong evidence of comparison between these techniques is available, especially for non-palpable BC lesions. To our knowledge, the only randomized clinical trial available analyzes the performances of IOUS only taking into consideration palpable lesions. Therefore, more robust randomized trials are needed in order to provide a complete picture of the real effectiveness of these new promising techniques.

The aim of this prospective trial is to identify which of these three techniques offers the best surgical guidance for non-palpable BC lesions excision in terms of surgical, oncological, cosmetic and cost-effectiveness outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-palpable breast cancer candidate for breast-conserving surgery;
* Female patients;
* Patients aged ≥ 18 years;
* Patients with histologic diagnosis of cT1-T2 invasive BC or ductal carcinoma in situ;
* Patients amenable for BCS after neoadjuvant chemotherapy;
* Patients who are able to give informed consent.

Exclusion Criteria:

* Pregnancy or lactation;
* Patients with locally advanced disease or metastatic disease;
* Patients with palpable breast carcinoma;
* Patients candidate for mastectomy;
* Patients who are unable to give informed consent
* Patients candidate for mastectomy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1302 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Involved resection margins. | Through study completion, an average of 2 years
  Compare the efficacy of the IOUS HydroMark™ and magnetic Sirius Pintuition Seed® versus the wire localization technique in terms of involved resection margins. Positive margin rate, defined as the number of patients with ink on invasive cancer or ductal carcinoma in situ with a resection margin < 2mm out of the total number of enrolled patients.

SECONDARY OUTCOMES:
Postoperative complications | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of postoperative complications, assessed according to the Clavien-Dindo classification system.
Re-excision rate | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of re-excision rate, defined as the number of patients who need to be re-operated after initial conservative surgery out of the total number of operated patients. Reoperation was recommended for any resection margin < 2 mm.
Target lesion removal rates | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of target lesion removal rates, defined as the number of lesions that were totally removed without involved margins after first surgical excision
Closest margin width | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of closest margin width, calculated as the minimal distance between the tumor edge and the closest resection margin
Calculated resection ratio (CRR) | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of calculated resection ratio (CRR), defined as the surgical specimen volume related to the optimal resection volume (ORV), which represent the theoretical minimum volume needed to remove the tumor with a 1 cm clear margin
Tumor and surgical specimen volume ratio | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of tumor and surgical specimen volume ratio: the tumor volume will be calculated considering the tumor as an elliptical sphere using the ellipsoid equation V = 4/3 pi × a × b × c, where a, b and c are the lengths of the semi-diameters of the tumor; the surgical specimen volume will be the sum of the main specimen and the cavity shaving margin volumes; these will be calculated as volumes of a rhombic prism, using the formula V = d1 × d2 × h/2, where d1, d2 and h are the diameters of the main specimen and of each single cavity shaving margin. Volumes that will be excised only for cosmetic reasons will not be considered.
BREAST-Q score | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of BREAST-Q score based on BREAST-Q BCT module, a questionnaire designed to evaluate patient satisfaction in two domains: satisfaction with breasts and satisfaction with care.
Resource consumption and estimation of costs | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of resource consumption and estimation of costs. Costs will be calculated in euros (€) for eachparticipant in the clinical trial. The economic evaluation is performed as a within-trial analysis, indicating that only costs and effects that accumulate within the trial length are included.
Number of re-excisions within the first 6 months following the first surgery | Through study completion, an average of 2 years
  Evaluate the 3 techniques in terms of number of re-excisions within the first 6 months following the first surgery.
EQ-5D-5L | Through study completion, an average of 2 years
  The patient-related effectiveness measures are health related quality of life (HRQoL). HRQoL is estimated using the EuroQol 5-dimension 5-level (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Ferrucci, MD PhD, Principal Investigator — Veneto Institute of Oncology IRCCS
Locations (5):
- Italy (5):
  - Azienda Ospedaliera San Giovanni Addolorata, Roma, RM
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - AOU Policlinico di Modena, Modena
  - ASL2 Abruzzo, Ospedale "Gaetano Bernabeo", Ortona, Ortona
  - Istituto Oncologico Veneto IRCCS, Padua

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krekel NM, Haloua MH, Lopes Cardozo AM, de Wit RH, Bosch AM, de Widt-Levert LM, Muller S, van der Veen H, Bergers E, de Lange de Klerk ES, Meijer S, van den Tol MP. Intraoperative ultrasound guidance for palpable breast cancer excision (COBALT trial): a multicentre, randomised controlled trial. Lancet Oncol. 2013 Jan;14(1):48-54. doi: 10.1016/S1470-2045(12)70527-2. Epub 2012 Dec 4. PMID 23218662
- [Background] Rubio IT, Esgueva-Colmenarejo A, Espinosa-Bravo M, Salazar JP, Miranda I, Peg V. Intraoperative Ultrasound-Guided Lumpectomy Versus Mammographic Wire Localization for Breast Cancer Patients After Neoadjuvant Treatment. Ann Surg Oncol. 2016 Jan;23(1):38-43. doi: 10.1245/s10434-015-4935-z. Epub 2015 Oct 29. PMID 26514120
- [Background] Volders JH, Haloua MH, Krekel NM, Negenborn VL, Kolk RH, Lopes Cardozo AM, Bosch AM, de Widt-Levert LM, van der Veen H, Rijna H, Taets van Amerongen AH, Jozwiak K, Meijer S, van den Tol MP. Intraoperative ultrasound guidance in breast-conserving surgery shows superiority in oncological outcome, long-term cosmetic and patient-reported outcomes: Final outcomes of a randomized controlled trial (COBALT). Eur J Surg Oncol. 2017 Apr;43(4):649-657. doi: 10.1016/j.ejso.2016.11.004. Epub 2016 Nov 23. PMID 27916314
- [Background] Esgueva A, Rodriguez-Revuelto R, Espinosa-Bravo M, Salazar JP, Rubio IT. Learning curves in intraoperative ultrasound guided surgery in breast cancer based on complete breast cancer excision and no need for second surgeries. Eur J Surg Oncol. 2019 Apr;45(4):578-583. doi: 10.1016/j.ejso.2019.01.017. Epub 2019 Feb 1. PMID 30737056
- [Background] Ferrucci M, Milardi F, Passeri D, Mpungu LF, Francavilla A, Cagol M, Saibene T, Michieletto S, Toffanin M, Del Bianco P, Grossi U, Marchet A. Intraoperative Ultrasound-Guided Conserving Surgery for Breast Cancer: No More Time for Blind Surgery. Ann Surg Oncol. 2023 Oct;30(10):6201-6214. doi: 10.1245/s10434-023-13900-x. Epub 2023 Aug 22. PMID 37606837